CLINICAL TRIAL: NCT01150669
Title: SCOR in Targeted Therapies for Infant Leukemia Project 3: Targeting FLT3 in Infant Leukemia
Brief Title: Lestaurtinib With or Without Chemotherapy Agents in Samples From Young Patients With Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML10B18; NCI-2011-02240 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-AAML10B18 (Other: Children's Oncology Group); CDR0000675724 (Other: Clinical Trials.gov)
Record Dates: First submitted 2010-06-24; First posted 2010-06-25 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Childhood Acute Lymphoblastic Leukemia; Childhood Acute Myeloid Leukemia/Other Myeloid Malignancies
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational: Cryopreserved specimens are studied in vitro with lestaurtinib with or without chemotherapy agents. Samples are analyzed for FLT3 protein expression and/or activation; sensitivity to lestaurtinib with or without chemotherapy agents; and activation of STAT, AKT, and RAS-MAPK and other pathways by western blot. The most effective treatment from this study is then validated in vivo in a NOD/SCID xenograft model.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Samples are analyzed in laboratory studies

SUMMARY:
This research study is studying lestaurtinib with or with chemotherapy in samples from young patients with leukemia. Studying the effects of lestaurtinib with or without chemotherapy in cell samples from patients with cancer in the laboratory may help doctors learn more about the effects of this treatment on cancer cells. It may also help doctors identify biomarkers related to cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the potential of lestaurtinib with or without chemotherapy agents in treating samples from infants with leukemia.

II. Determine whether FLT3 protein expression level and/or activation and sensitivity to lestaurtinib differ between subgroups of infants with leukemia.

III. Determine whether lestaurtinib activates STAT5, AKT, and RAS-MAPK and other pathways.

IV. Determine whether lestaurtinib can synergize with other chemotherapy agents kill infant leukemia cells.

OUTLINE: This is a multicenter study.

Cryopreserved specimens are studied in vitro with lestaurtinib with or without chemotherapy agents. Samples are analyzed for FLT3 protein expression and/or activation; sensitivity to lestaurtinib with or without chemotherapy agents; and activation of STAT, AKT, and RAS-MAPK and other pathways by western blot. The most effective treatment from this study is then validated in vivo in a NOD/SCID xenograft model.

ELIGIBILITY:
Inclusion Criteria:

* Cryopreserved samples from infants with leukemia available

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Samples from infants with leukemia
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2010-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Expression level and activation state of FLT3 protein, determined by Western blotting and FACS | Up to 4 months
TKI sensitivity, determined by MTT and annexin V assays | Up to 4 months
Baseline activation and inhibition of STAT5, AKT, and RAS-MAPK and other pathways, examined with Western blotting and phosphospecific antibodies | Baseline
Incidence of cell death in primary infant leukemia samples treated with sequenced combinations of chemotherapy and FLT3 TKI using MTT and annexin V binding assays and median effect analysis | Up to 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Brown, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Monrovia, California, United States